CLINICAL TRIAL: NCT01351779
Title: The Effect of Body Posture on Intraocular Pressure in Progressive Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Sensimed AG (Industry)
Responsible Party: Professor Graham Trope, University of Toronto
Other Study IDs: 10-0844-A
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Glaucoma
Keywords: Intraocular pressure; Contact lens sensor; Optic disc hemorrhage
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Progressive glaucoma: Patients with primary open angle glaucoma identified to have an optic disc hemorrhage

SUMMARY:
Glaucoma is a condition where the optic nerve (the nerve responsible for sight) shows progressive damage with characteristic loss of visual field. Glaucoma is very commonly associated with raised pressure in the eye (intraocular pressure [IOP]). IOP has been shown to increase when lying down in normal subjects as well as patients with glaucoma. It is possible that this effect can make glaucoma worse. This study is designed to investigate the effect of body posture (particularly when sleeping) on the IOP fluctuation in the eye. Each patient will be required to attend for 2 separate 24 hour visits. On one visit the patient will be required to sleep flat and on the other visit at a 30° head up sleeping position. During this time the patient will be required to wear a soft contact lens (SENSIMED Triggerfish®) which has a special sensor on it that monitors the IOP continuously. The IOP measurements are wirelessly transmitted to a recorder.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* diagnosis of primary open angle glaucoma (POAG) or normal tension glaucoma (NTG) that is progressing based on recent or recurrent optic disc hemorrhage
* age 18-85 years
* not more than 4 diopters of spherical equivalent or 2 diopters of cylinder equivalent in study eye
* stable anti-glaucoma treatment for 4 weeks before first session
* for women of childbearing potential, adequate contraception

Exclusion Criteria:

* unwilling or unable to sleep in a flat or 30 degrees head up position
* ocular surgery in previous 3 months
* corneal or conjunctival abnormality
* wear of full frame metallic glasses during monitoring session
* severe dry eye
* secondary forms of glaucoma
* allergy to corneal anaesthesia
* patients with contraindications for contact lens wear
* pregnancy and lactation
* patients unable to understand the character and individual consequences of the investigation
* simultaneous participation in other research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure changes that occur during sleep and with changes in body posture | 24 hours
  The intraocular pressure will be continuously monitored with a wireless contact lens sensor device over a 24 hour period

SECONDARY OUTCOMES:
Incidence of side effects or adverse effects that occur while subjects are wearing the contact lens device | 24 hours
  Patients will be monitored for contact lens related side effects or adverse effects that occur during the monitoring session.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Beltran-Agullo L, Buys YM, Jahan F, Shapiro CM, Flanagan JG, Cheng J, Trope GE. Twenty-four hour intraocular pressure monitoring with the SENSIMED Triggerfish contact lens: effect of body posture during sleep. Br J Ophthalmol. 2017 Oct;101(10):1323-1328. doi: 10.1136/bjophthalmol-2016-308710. Epub 2017 Mar 7. PMID 28270491